CLINICAL TRIAL: NCT03447587
Title: Determining the Role of Acupuncture in the Modulation of Peripheral Oxidative Stress in Patients With Insomnia: A Randomized Placebo-Controlled Trial
Brief Title: Acupuncture in the Modulation of Peripheral Oxidative Stress Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, YEUNG Wing Fai, Assistant professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AcupOS
Record Dates: First submitted 2018-01-17; First posted 2018-02-27 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Insomnia Chronic
Keywords: Randomized controlled trial; Sleep; Traditional Chinese medicine; Oxidative stress
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: Randomized to two groups in 1:1 ratio.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture (Experimental): Subjects will receive 4 weeks of acupuncture following with a semi-standardized protocol.
  Interventions: Other: Electroacupuncture
- Sham acupuncture group (Placebo Comparator): Subjects will receive sham acupuncture with the same sterilization procedure as traditional acupuncture group.
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: Electroacupuncture — Each subject will be treated with predefined acupoints including bilateral Ear-Shenmen, Touwei (ST8), Sishencong (EX-HN1), and unilateral Yintang (EXHN3) and Baihui (GV20) on the head (total 8 needles). Subject's current symptoms will be ascertained using a Traditional Chinese Medicine symptom checklist and eight additional acupoints will therefore be selected and needled based on their clinical judgements. The acupuncture treatment will consistent of two sessions per week (30 minutes) for 4 consecutive weeks.
  Arms: Electroacupuncture
Other: Sham acupuncture — Subjects will be treated at 1 cm posteriorly and laterally adjacent to the same acupoints as the traditional acupuncture group using validated non-invasive sham needles. Subjects will also be assessed with Traditional Chinese Medicine checklist. The acupuncturist, setting, treatment frequency, and duration of the treatment course will be the same as in the traditional acupuncture group.
  Arms: Sham acupuncture group

SUMMARY:
A randomized controlled trial involving 140 subjects with (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) DSM-5 insomnia disorder after excluding those with other medical conditions, psychiatric disorders, and sleep disorders that may cause insomnia. The subjects will be randomly assigned to either acupuncture treatment or sham acupuncture (control group) in a 1:1 ratio. The acupuncture treatment group will receive acupuncture treatments using a semi-standardized protocol. In a similar way, the sham acupuncture control group will receive acupuncture using validated non-invasive sham acupuncture needles. Both subjective (the sleep questionnaire and sleep diary) and objective (actigraphy) outcome measures will be recorded at baseline and at 1- and 5-week post-treatment. Fasting blood samples will be taken on the morning of the assessments at these time points to measure the oxidative stress parameters, including the malondialdehyde (MDA) level, and the glutathione peroxidase (GPx), paraoxonase (PON), and arylesterase (ARE) activities. The primary outcome is sleep efficiency, measured using a 7-day sleep diary and the oxidative stress parameters at 1-week post-treatment.

DETAILED DESCRIPTION:
Background: Insomnia is a very common complaint worldwide. Acupuncture is an alternative treatment for improving sleep quality. However, its efficacy and mechanism of action as a treatment for insomnia requires further investigation. Acupuncture may attenuate oxidative stress which is thought to be an important pathophysiological factor in insomnia.

Aims: To evaluate the safety and efficacy of a semi-individualized acupuncture treatment in improving sleep, and to examine its effects on oxidative stress parameters in subjects with primary insomnia disorder.

Methods: This will be a randomized controlled trial involving 140 subjects with DSM-5 insomnia disorder after excluding those with other medical conditions, psychiatric disorders, and sleep disorders that may cause insomnia. The subjects will be randomly assigned to either acupuncture treatment or sham acupuncture (control group) in a 1:1 ratio. The acupuncture treatment group will receive acupuncture treatments using a semi-standardized protocol. In a similar way, the sham acupuncture control group will receive acupuncture using validated non-invasive sham acupuncture needles. Both subjective (the sleep questionnaire and sleep diary) and objective (actigraphy) outcome measures will be recorded at baseline and at 1- and 5-week post-treatment. Fasting blood samples will be taken on the morning of the assessments at these time points to measure the oxidative stress parameters, including the malondialdehyde (MDA) level, and the glutathione peroxidase (GPx), paraoxonase (PON), and arylesterase (ARE) activities. The primary outcome is sleep efficiency, measured using a 7-day sleep diary and the oxidative stress parameters at 1-week post-treatment.

Data analysis: Changes in the sleep and oxidative stress outcome measures will be compared between groups by using a mixed-effects model at each time point. Correlations between sleep parameters and oxidative stress parameters will be examined using a Pearson correlation. Mediation analysis will be performed to explore the possible mediating effect of oxidative stress factors on sleep.

Significance: The relationship between oxidative stress and insomnia severity has been under-researched. To the best of our knowledge, there has thus far been no study on the effect of acupuncture on oxidative stress in subjects with insomnia disorder. The present study will not only provide high-quality evidence of the efficacy of acupuncture as a treatment for insomnia, but also of the associated changes in oxidative stress parameters. It will guide future studies on the treatment mechanism and pathophysiology of insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong resident,
* ethnic Hong Kong Chinese aged 18-65,
* fulfilling diagnostic criteria of insomnia disorder using DSM-5 diagnostic criteria for Insomnia Disorder by Brief Insomnia Questionnaire,
* Insomnia Severity Index total score ≥11 at screening and baseline visits,
* willing to give informed consent and comply with the trial pr1otocol.

Exclusion Criteria:

* any current or past major depressive disorder, generalized anxiety disorders or panic disorder, manic or hypomanic episode, substance use disorders, organic mental disorder, schizophrenia or any other psychotic disorder as defined by DSM-IV criteria using the Structured Clinical Interview for DSM-IV (SCID);
* any current physical illnesses that contributes significantly to the subject's insomnia;
* pregnancy;
* a previous diagnosis of sleep apnea or periodic limb movement disorder (if subjects with symptoms suggestive of other sleep disorders, they will be referred to our psychiatrists for further assessment;
* a Home Single-Channel Nasal Pressure (HNP) screening with apnea-hypopnea index (AHI) >5;
* at significant risk of suicide according to SCID;
* infection or abscess close to the site of the selected acupoints;
* valvular heart defects, bleeding disorders or taking anticoagulant drugs, use of any implanted electrical device such as pacemaker, defibrillator, brain and nerve stimulators, etc.;
* receiving acupuncture treatment in the past 6 months;
* taking herbal remedies, over-the-counter medication or psychotropic drugs that target insomnia within the two weeks prior to baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency (SE) | Week 5
  the sleep efficiency derived from 7 days sleep diary

SECONDARY OUTCOMES:
Sleep efficiency (SE) | Baseline, week 9
  the sleep efficiency derived from 7 days sleep diary
Sleep onset latency (SOL) | Baseline, week 5, week 9
  the sleep onset latency derived from 7 days sleep diary
Wake after sleep onset (WASO) | Baseline, week 5, week 9
  the Wake after sleep onset derived from 7 days sleep diary
Total sleep time (TST) | Baseline, week 5, week 9
  the total sleep time derived from 7 days sleep diary
Insomnia Severity Index (ISI) | Baseline, week 5, week 9
  the self reported severity of insomnia symptoms
Hospital Anxiety and Depression (HADS) | Baseline, week 5, week 9
  the self reported anxiety and depression symptoms
Short Form Six Dimension (SF6D) | Baseline, week 5, week 9
  the six dimension measure of health-related quality of life
Actigraphy: Sleep onset latency (SOL) | Baseline, week 5, week 9
  The objective measure of sleep onset latency (SOL)
Actigraphy: Wake after sleep onset (WASO) | Baseline, week 5, week 9
  The objective measure of wake after sleep onset (WASO)
Actigraphy: Total sleep time (TST) | Baseline, week 5, week 9
  The objective measure of total sleep time (TST)
Actigraphy: Sleep efficiency (SE) | Baseline, week 5, week 9
  The objective measure of sleep efficiency (SE)
The level of MDA | Baseline, week 5
  The measure of oxidative stress parameters
The activity of GPx | Baseline, week 5
  The measure of oxidative stress parameters
The activity of PON | Baseline, week 5
  The measure of oxidative stress parameters
The activity of ARE | Baseline, week 5
  The measure of oxidative stress parameters

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, the Hong Kong Polytechnic University, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Yeung WF, Yu BY, Yuen JW, Ho JYS, Chung KF, Zhang ZJ, Mak DSY, Suen LK, Ho LM. Semi-Individualized Acupuncture for Insomnia Disorder and Oxidative Stress: A Randomized, Double-Blind, Sham-Controlled Trial. Nat Sci Sleep. 2021 Jul 21;13:1195-1207. doi: 10.2147/NSS.S318874. eCollection 2021. PMID 34321944